CLINICAL TRIAL: NCT03559231
Title: Endoscopic Resection of Non-ampullary Duodenal Adenomas: Endoscopic Mucosal Resection (EMR) vs. Endoscopic Full-thickness Resection With the 'Duodenal Full-thickness Resection Device' (dFTRD)
Acronym: DUO-RESECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kliniken Ludwigsburg-Bietigheim gGmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DUO-RESECT
Record Dates: First submitted 2018-05-11; First posted 2018-06-18 (Actual); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Duodenal Adenoma
Keywords: duodenal adenoma; FTRD; dFTRD; EMR; endoscopic mucosal resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dFTRD (Experimental): Endoscopic full-thickness resection of the duodenal adenoma with the 'duodenal Full-Thickness resection device' (dFTRD).
  Interventions: Procedure: dFTRD
- EMR (Active Comparator): Endoscopic Mucosal Resection (EMR) of the duodenal adenoma (=standard therapy).
  Interventions: Procedure: EMR

INTERVENTIONS:
Procedure: dFTRD — Duodenal Full-Thickness Resection
  Arms: dFTRD
Procedure: EMR — Endoscopic Mucosal Resection
  Arms: EMR

SUMMARY:
Prospective, randomized multi-center trial. Comparison of Endoscopic Mucosal Resection (EMR) versus Endoscopic Full-Thickness Resection with the duodenal Full-Thickness Resection Device (dFTRD) of non-ampullary duodenal adenomas.

DETAILED DESCRIPTION:
Prospective, randomized multi-center trial. Comparison of Endoscopic Mucosal Resection (EMR) versus Endoscopic Full-Thickness Resection with the duodenal Full-Thickness Resection Device (dFTRD) of non-ampullary duodenal adenomas.

ELIGIBILITY:
Inclusion Criteria:

* duodenal adenoma
* age 18 or older
* written informed consent

Exclusion Criteria:

* duodenal adenomas with a size > 25 mm
* duodenal adenomas with 20 mm or less distance to the major and/or minor duodenal papilla
* presence of two or more duodenal adenomas
* suspected or histologically confirmed malignancy
* tumor disease (exception: after successful curative treatment)
* conditions/diseases of the upper GI-tract that impair advancing of the devices into the duodenum
* moribund patient
* pregnancy and breastfeeding
* patients that cannot give informed consent (e.g. psychiatric disorders, language barrier,...)
* other contraindications for duodenal resections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-05-12 (Actual); Primary Completion 2020-06-12 (Estimated); Study Completion 2021-05-12 (Estimated)

PRIMARY OUTCOMES:
Complication Rate | 30 days
  Composite endpoint of perforations and relevant bleeding

SECONDARY OUTCOMES:
Technical success | intraoperative
  Rate of macroscopic complete resections
'R0'-Resection | within one week after resection (as soon as result of pathologic analysis of resected specimen is available)
  Rate of microscopic complete resections
Rate of 'en bloc' resections | within one week after resection (as soon as result of pathologic analysis of resected specimen is available)
  Rate of 'en bloc' resections
Need of secondary surgical intervention | 3 months
Procedure time | 30 days
  time span of the procedure according to sedation protocol
Duration of hospitalization | 30 days
number of patients with residual or recurrent duodenal adenoma at the follow-up endoscopy after 3 months | 3 months
number of patients with residual or recurrent duodenal adenoma at the follow-up endoscopy after 1 year | 1 year
number of necessary re-endoscopies | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Karel Caca, MD, PhD, Study Chair — Klinikum Ludwigsburg
Locations (1):
- Klinikum Ludwigsburg, Ludwigsburg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No